CLINICAL TRIAL: NCT06434792
Title: A Multicenter, Randomized, Double-blind, Placebo-controlled, Parallel-group Dose-response Phase 2 Clinical Trial to Compare the Efficacy and Safety of Bronpass Tab. Versus Placebo in Patients With Stable COPD
Brief Title: Study to Evaluate Efficacy and Safety of Bronpass Tab. in Patients With Chronic Obstructive Pulmonary Disease
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Hanlim Pharm. Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: HL_HL301_204
Record Dates: First submitted 2023-09-18; First posted 2024-05-30 (Actual); Last update posted 2024-05-30 (Actual); Status verified 2024-05

CONDITIONS: Chronic Obstructive Pulmonary Disease
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Bronpass Tab. (Experimental): Twice daily for 12 weeks
  Interventions: Drug: Bronpass Tab.
- Placebo (Placebo Comparator): Twice daily for 12 weeks
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Bronpass Tab. — Twice daily for 12 weeks
  Other Names: HL301
  Arms: Bronpass Tab.
Other: Placebo — Twice daily for 12 weeks
  Arms: Placebo

SUMMARY:
This clinical trial is a multicenter, randomized, double-blind, placebo-controlled, parallel-group dose-response phase 2 clinical trial study to evaluate the efficacy and safety of Bronpass Tab. in 96 patients with chronic obstructive pulmonary disease.

DETAILED DESCRIPTION:
This study is to prove that Bronpass Tab. is superior in clinical efficacy and safety in improving COPD symptoms compared to placebo for 12 weeks in patients suffering from chronic obstructive pulmonary disease.

ELIGIBILITY:
Inclusion Criteria:

1. 40 years ≤ age
2. Patients who are diagnosed as COPD (based on the definition in the Korean Society of Tuberculosis and Respiratory Diseases COPD Guidelines)
3. Patients who meet all of the following criteria at the screening test

   * FEV1/FVC < 0.70 after bronchodilator administration
   * 30% ≤ FEV1 < 80% predicted after bronchodilator administration
   * Cough or sputum-related score on the CAT ≥ 3
4. Current or former smokers with a smoking history of 10 pack-years or more at screening.
5. Patients who have listened to a detailed explanation of this clinical trial, fully understand it, and voluntarily provide written consent to participate.

Exclusion Criteria:

1. Patients with a current medical history of asthma (However, patients previously diagnosed as asthma who have recovered and currently have a diagnosis of COPD are eligible for participation.)
2. Patients with a medical history of respiratory diseases other than COPD
3. Patients who have undergone lung volume reduction surgery.
4. Patients with a history of lung transplantation.
5. Patients with a history of respiratory infections within 4 weeks prior to screening
6. Patients with a history of moderate or severe acute exacerbation within 4 weeks prior to screening.
7. Pregnant or lactating women.
8. Patients who are considered ineligible for this clinical trial due to other reasons as judged by the investigator.

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 96 (Estimated)
Dates: Start 2023-06-01 (Actual); Primary Completion 2024-09 (Estimated); Study Completion 2025-03 (Estimated)

PRIMARY OUTCOMES:
Change from baseline in CAT(COPD Assessment Test) total score at Visit 5 | Time frame: 3 months(Visit 5)

SECONDARY OUTCOMES:
Change from baseline in CAT total score at Visit 3 and Visit 4 | Time frame: 1 month(Visit 3), 2 months(Visit 4)
Change from baseline in CAT cough score at Visit 3, Visit 4, and Visit 5 | Time frame: 1 month(Visit 3), 2 months(Visit 4), 3 months(Visit 5)
Change from baseline in CAT sputum score at Visit 3, Visit 4, and Visit 5 | Time frame: 1 month(Visit 3), 2 months(Visit 4), 3 months(Visit 5)
Incidence of moderate and severe COPD exacerbations from baseline to Visit 5 | Time frame: 3 months(Visit 5)
Change frome baseline in PFT(Pulmonary Function Test) such as FEV1(Forced Expiratory Volume in one second), FVC(Forced Vital Capacity), FEV1/FVC at Visit 5 | Time frame: 3 months(Visit 5)
Change from baseline in SGRQ-C(St. George's Respiratory Questionnaire for COPD patients) Score at Visit 3, Visit 4, and Visit 5 | Time frame: 1 month(Visit 3), 2 months(Visit 4), 3 months(Visit 5)
Change from baseline in COAT(Cough Assessment Test) Score at Visit 3, Visit 4, and Visit 5 | Time frame: 1 month(Visit 3), 2 months(Visit 4), 3 months(Visit 5)

CONTACTS AND LOCATIONS:
Overall Officials: Kwang Ha Yoo, MD, PhD, Principal Investigator — Konkuk University
Locations (1):
- Konkuk University School of Medicine, Seoul, South Korea